CLINICAL TRIAL: NCT03915249
Title: Investigation of Relationship Among Physical Activity, Pulmonary Functions and Physical Functions in Candidates With Allogeneic Hematopoietic Stem Cell Transplantation: a Cross Sectional Study
Brief Title: Physical Functions in Allogeneic-HSCT Candidates
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Associate professor, Gazi University
Other Study IDs: GaziUniversity17
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Stem Cell Transplantation
Keywords: Energy metabolism; Exercise test; Leisure activities; Hematopoietic stem cell transplantation; Muscle strength; Respiratory function test; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allogeneic-HSCT candidates: Physical activity, pulmonary functions (FEV1, FVC, FEV1/FVC, FEF25-75%, PEF), exercise capacity, respiratory (maximal inspiratory and expiratory pressures (MIP, MEP)) and peripheral muscle strength were evaluated in allogeneic-HSCT candidates.

SUMMARY:
Physical inactivity and impairments in physical functions have been observed in patients due to hematological malignancy itself and treatments of chemotherapy, radiotherapy, corticosteroids. However, no study investigated relationship of physical activity with pulmonary and physical functions in allogeneic hematopoietic stem cell transplantation (HSCT) candidates. Therefore, investigation of the relationship among outcomes in allogeneic HSCT candidates was aimed.

DETAILED DESCRIPTION:
Hematological malignancies arise from deficiencies in blood cell lineage which represent a heterogeneous group including leukemias, lymphomas, myelomas, myeloproliferative diseases and myelodysplastic syndromes. In recent years, a great majority of patients with hematological malignancies often experience side effects of disease related treatments such as chemotherapy with multiple agents, radiotherapy, corticosteroids, combination of medical drugs, autologous and/or allogeneic hematopoietic stem cell transplantation (HSCT) throughout their remaining lives. Furthermore, there are substantial outcomes regarding the initial time of diagnosis that pulmonary function involvements, sedentary life style (39%), decreased exercise capacity and lower extremity muscle weakness have been present in patients with lymphoma even before first cycle of chemotherapy is administered to patients. During the period of or after chemotherapy, patients have suffered from decreased maximal oxygen uptake, advanced muscle weakness, decreased hemoglobin levels and evident fatigue, as well.

As the treatment process continues for patients with hematological malignancies, HSCT is begun to schedule for almost all patients which has a significant potential for good clinical outcomes along with longer life expectancy. However, especially allogeneic-HSCT is a quite aggressive treatment option due to serious complications such as graft versus host disease, long term severe treatments of these complications and severe immune suppression related infections. Moreover, patients have already been exposed to immobility condition, low level of physical activity, pulmonary functions involvements, respiratory and peripheral muscle weakness as well as exercise intolerance before HSCT. In addition, the outcomes obtained from candidates just before HSCT have indicated that quadriceps femoris muscle strength, exercise capacity evaluated with 6-minute walk test, inspiratory and expiratory muscle strength are decreased respectively in 23%, 58%, 42% and 89% of candidates. Sarcopenia (50.6%), reduction in hip flexor, hip abductors and ankle flexors muscles strength and decreased diffusing capacity of the lung for carbon monoxide (78%) have also been mostly observed in HSCT candidates. In a study, candidates who were evaluated using a metabolic holter device are inactive (average 2180 steps/day) before HSCT. In another study, number of steps evaluated using a pedometer which provides only one output about step count are approximately 201.1 steps per a day for HSCT candidates. Accuracy of pedometers can be reduced at slow walking speeds so that pedometers may not be suitable for cancer patients. On the other hand, metabolic holter devices use pattern recognition technology to evaluate physical activity level that may produce more accurate estimation of energy expenditure in cancer population. Besides, it has also been stated that quadriceps femoris muscle weakness is related to reduced daily number of steps, therefore if the muscles are strengthened, number of steps may be increased at the process of HSCT.

Physical activity is any bodily movement which is produced by skeletal muscles concluded energy expenditure. While total daily energy expenditure demonstrates all types of energy costs including resting, diet-induced and activity-induced energy expenditures within 24 hours, active energy expenditure related with physical activity is produced by daily living activities such as employment, sport and any other activities. Activity energy expenditure also decreases with excess body weight, older age, female gender, loss of muscle mass and diseases throughout life span . On the other hand, Canadian Academy of Sports and Exercise Medicine recommends that people prefer moderate-to-vigorous physical activity (>3.0 metabolic equivalents (METs)) including brisk walking, aerobic and resistance exercises, jogging, hiking, swimming and field games with ball or racquet for 150 min/week and a total sustainable activity duration from 30 min to 60 min per practice rather than sedentary behavior (<1.5 METs) in order to decrease risk of most major chronic disease by 25-50%. Moreover, a 15 min/d or 75 min/week of moderate-to-vigorous physical activity is also recommended as about 15% mortality risk reduces in diseases and benefits increase . Given the importance of physical activity assessment and counseling in people with/without chronic disease, according to literature, studies objectively investigating either detailed physical activity condition rather than number of steps or relations of physical activity with pulmonary and physical functions in allogeneic-HSCT candidates are scarce. Therefore, primary aim of the current study was to exhibit possible all detailed aspects of physical activity outcomes evaluated with a metabolic holter, an objective measurement device, secondary aim was to investigate relationship among physical activity parameters, pulmonary functions and physical functions in allogeneic-HSCT candidates and as finally, to identify independent predictors of physical inactivity in candidates was aimed.

ELIGIBILITY:
Inclusion Criteria:

* being 18-65 years of age,
* having a diagnosis with hematologic malignancy
* being clinically stabile,
* being an allogeneic-HSCT candidate
* receiving optimal standard medical therapy including antibiotics, supplements and other drugs.

Exclusion Criteria:

* having cooperation problems,
* having orthopedic or neurological disease with a potential to prevent assessment of exercise capacity,
* having comorbidities such as chronic obstructive pulmonary disease, cardiac diseases,
* acute infections and/or hemorrhage.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients were previously diagnosed with a hematological malignancy and determined to be a candidate for allogeneic-HSCT who were orientated from Bone Marrow Transplantation Unit for rehabilitation program.Study was planned as retrospective, cross sectional and approved by the local Ethics Committee. Informed consent was obtained from all individual participants included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Physical activity measurement | during a total of 48 hours
  Physical activity levels of candidates were assessed with a metabolic holter device.

SECONDARY OUTCOMES:
Pulmonary function assessment | 5 minutes
  It was evaluated using a spirometry by which is evaluated dynamic lung functions involving forced vital capacity (FVC), forced expiratory volume in one second (FEV1), forced expiratory volume in one second/forced vital capacity (FEV1/FVC), peak expiratory flow (PEF) and forced expiratory flow at 25%-75% (FEF25-75%). All of them are expressed as both liter (L) and percentages (%) of expected values. We used only percentages (%) of expected values for this study.
inspiratory and expiratory muscle strength (MIP, MEP) | 5-10 minutes
  Respiratory muscle strength was evaluated with a mouth pressure device
Quadriceps femoris muscle strength | 5 minutes
  Peripheral muscle strength was evaluated with a hand-held dynamometer
Six-minute walk test | 10 minutes
  Six-minute walk test was used to evaluate exercise capacity of candidates with reference to American Thoracic Society criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Barğı, PhD, Study Chair — Gazi University; Meral Boşnak Güçlü, PhD, Study Director — Gazi University; Gülsan Türköz Sucak, PhD., Principal Investigator — Medikalpark hastanesi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bergenthal N, Will A, Streckmann F, Wolkewitz KD, Monsef I, Engert A, Elter T, Skoetz N. Aerobic physical exercise for adult patients with haematological malignancies. Cochrane Database Syst Rev. 2014 Nov 11;(11):CD009075. doi: 10.1002/14651858.CD009075.pub2. PMID 25386666
- [Result] Vermaete N, Wolter P, Verhoef G, Gosselink R. Physical activity and physical fitness in lymphoma patients before, during, and after chemotherapy: a prospective longitudinal study. Ann Hematol. 2014 Mar;93(3):411-24. doi: 10.1007/s00277-013-1881-3. Epub 2013 Aug 21. PMID 23963412
- [Result] Gillis TA, Donovan ES. Rehabilitation following bone marrow transplantation. Cancer. 2001 Aug 15;92(4 Suppl):998-1007. doi: 10.1002/1097-0142(20010815)92:4+3.0.co;2-k. PMID 11519026
- [Result] Steinberg A, Asher A, Bailey C, Fu JB. The role of physical rehabilitation in stem cell transplantation patients. Support Care Cancer. 2015 Aug;23(8):2447-60. doi: 10.1007/s00520-015-2744-3. Epub 2015 May 14. PMID 25971213
- [Result] Hung YC, Bauer J, Horsley P, Waterhouse M, Bashford J, Isenring E. Changes in nutritional status, body composition, quality of life, and physical activity levels of cancer patients undergoing autologous peripheral blood stem cell transplantation. Support Care Cancer. 2013 Jun;21(6):1579-86. doi: 10.1007/s00520-012-1698-y. Epub 2013 Jan 10. PMID 23306934
- [Result] White AC, Terrin N, Miller KB, Ryan HF. Impaired respiratory and skeletal muscle strength in patients prior to hematopoietic stem-cell transplantation. Chest. 2005 Jul;128(1):145-52. doi: 10.1378/chest.128.1.145. PMID 16002928
- [Result] Morishita S, Kaida K, Ikegame K, Yoshihara S, Taniguchi K, Okada M, Kodama N, Ogawa H, Domen K. Impaired physiological function and health-related QOL in patients before hematopoietic stem-cell transplantation. Support Care Cancer. 2012 Apr;20(4):821-9. doi: 10.1007/s00520-011-1156-2. Epub 2011 Apr 9. PMID 21479522